CLINICAL TRIAL: NCT04649619
Title: Roux-en-Y Gastric Bypass as a Therapeutic Option for Patients With Indication for Bariatric and / or Metabolic Surgery: Clinical Trial
Brief Title: Roux-en-Y Gastric Bypass: Clinical Trial
Acronym: ERAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paulo Reis Esselin de Melo (Other)
Collaborators: Hospital Estadual Geral de Goiânia Dr. Alberto Rassi (Unknown)
Responsible Party: Sponsor-Investigator, Paulo Reis Esselin de Melo, Principal Investigator, Instituto Paulo Reis
Organization: Instituto Paulo Reis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UTN - U111112498106
Record Dates: First submitted 2020-08-07; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Anastomosis, Roux-en-Y; Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Prospective clinical trial with intentional sample selection that aims to describe the results of the gastric bypass surgery modified by De Melo, for the purpose of endoscopic access to the excluded remaining stomach, as well as to monitor the clinical conditions of comorbidities and the patient's quality of life.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm-study (Other): Prospective clinical trial with intentional sample selection that aims to describe the results of the gastric Bypass surgery modified by De Melo, for the purpose of endoscopic access to the excluded remaining stomach, as well as to monitor the clinical conditions of comorbidities and the quality of life of the patient.
  Interventions: Procedure: GASTRIC BYPASS MODIFIED IN ROUX-EN-Y AS A THERAPEUTIC OPTION IN PATIENTS WITH INDICATION OF BARIATRIC AND / OR METABOLIC SURGERY

INTERVENTIONS:
Procedure: GASTRIC BYPASS MODIFIED IN ROUX-EN-Y AS A THERAPEUTIC OPTION IN PATIENTS WITH INDICATION OF BARIATRIC AND / OR METABOLIC SURGERY — Roux-en-Y gastric bypass:
  Stapling and reduction of the gastric chamber of approximately 18 cm, followed by anastomosis with a deviated bowel, and another bowel anastomosis with a bowel in a lower portion, for deviation of biliopancreatic secretions. Maintenance of a gastro-gastric communication of approximately 1 cm between the functional gastric pouch and the excluded stomach for endoscopic access.
  Other Names: ROUX-EN-Y MODIFIED GASTRIC BYPASS

SUMMARY:
The present study aims to describe the results of a modified gastric bypass surgery to ensure endoscopic access to the excluded remaining stomach, as well as to monitor the clinical conditions of comorbidities and the patient's quality of life, since associated complications can be found to the excluded stomach, such as: bile reflux, gastritis and / or gastric and duodenal ulcer, H. pylori infection, bleeding, gastric polyps and the possibility of gastric cancer in patients undergoing RYGB (Roux-en-Y gastric bypass), with one of the probable factors being the occurrence reflux of the duodenal content into the excluded portion of the stomach.

In this sense, based on technical concepts of an established surgical procedure, the RYGB, the present project is not a proposal for a new procedure, but an adaptation of an existing technique. The proposal of the present study is about adaptations in RYGB surgery, which will enable endoscopic access to the remaining stomach, through the creation of a gastric communication.

DETAILED DESCRIPTION:
This is a prospective clinical trial with intentional sample selection, which will last 18 months and will be developed at the General State Hospital of Goiânia Alberto Rassi (HGG).

The present study aims at gastric bypass surgery modified for the purpose of ensuring endoscopic access to the excluded remaining stomach, as well as monitoring the clinical conditions of comorbidities and the patient's quality of life; evaluating the loss of excess body weight of 50% (EBW50%), as recommended by the World Health Organization and the Brazilian Society of Bariatric and Metabolic Surgery, to comparing weight loss before and after surgery; comparing the incidence and control of comorbidities associated with excess body weight, if the patient has any, before and after the surgery analyzing the nutritional characteristics of the patients before and after the surgery and its relationship with the obesity of their comorbidities; evaluating and comparing patients' quality of life before and after bariatric surgery;measuring and comparing lung function, respiratory muscle strength and endurance, physical fitness and functional capacity. The estimated sample size was calculated in the Epi Info Software (version 7.2.3.1) considering a 95% Confidence Interval, average volume of bariatric surgeries performed in the last year at HGG (p = 288) and an occurrence of bile reflux after RYGB 1.9%. When considering an estimated margin of error of 5%, the total value of twenty-six patients was found to compose the sample.

Predicting the occurrence of possible losses from follow-up throughout the study, a margin of 30% was added to the calculated value, ending with a total of 33 patients to compose the sample. Free-demand patients at the State Hospital of Goiânia Alberto Rassi, who have an indication for bariatric and / or metabolic surgery confirmed by the medical and multidisciplinary team, will be selected as potential participants in the research. The patient will be invited to participate in the study, receiving complete information about the planned procedures, risks and possible benefits.

The patient's refusal to participate in the research will not result in discontinuation of treatment. The baseline clinical parameters of the selected patients (age, weight, BMI, blood pressure, presented comorbidities, cardiovascular history, previous clinical treatments for the control of DM2 (Type 2 diabetes Mellitus), eating habits and physical activity) will be collected and inserted in clinical records during preoperative multidisciplinary consultation.

Data on food consumption will be collected in the preoperative period and in the postoperative period of 6, 12 and 18 months, through the application of the Food Frequency questionnaire.

In addition to collecting this information, the patient will be referred for preoperative exams, which will also be recorded in the patient's medical record. After fulfilling the criteria and after signing the Informed Consent Form, thirty-three patients will be selected who meet the inclusion and exclusion criteria to perform the modified RYGB technique to maintain gastro-gastric communication for endoscopic study after surgery.

Patients will undergo a consultation with the multidisciplinary team, when they will receive nutritional, psychological and physiotherapy team guidance. Once the date of the surgery is scheduled, the participants must follow the following regimen: absolute fasting of 8 hours before surgery, prophylactic dose of anticoagulant 12 hours before the surgery. Patients will be admitted 24 to 48 hours before the surgical procedure.

The surgery will be performed at the General State Hospital of Goiânia Alberto Rassi. After the preoperative procedure, the patient will be submitted to general anesthesia. Prophylactically, the patient will receive a single dose of 2 to 3 grams of kefazol 1 hour before the procedure, and to allergies 600 to 900 mg of intravenous clindamycin, and pneumatic socks and leggings will be provided to prevent thromboembolic events. For safety reasons, the patient will be monitored throughout the surgical procedure using multiparametric electronic monitors and bladder catheterization.

Initially, a median laparotomy will be performed with the measurement of the length of the entire small intestine, followed by an approach to the small curvature of the stomach, where it will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes;
* Minimum age of 18 and maximum of 70 years for a BMI greater than or equal to 35 kg / m2;
* Age from 30 to 70 years for BMI greater than or equal to 30 and less than or equal to 34.9 kg / m2, associated with diabetes;
* Absence of contraindications for the surgical procedure.

Exclusion Criteria:

* Abandonment of pre-operative multiprofessional follow-up before 12 months;
* Members of vulnerable groups;
* Uncompensated psychiatric disorders or cognitive impairment confirmed by a psychiatrist and / or psychologist;
* Abuse of alcohol or illicit drugs confirmed after evaluation by the psychiatrist and / or psychologist;
* Chronic diseases not related to obesity such as cancer, pneumopathy, nephropathy, heart disease, Parkinson's and Alzheimer's.
* Patients already undergoing other bariatric surgeries.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-01-18 (Actual); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-04-29 (Estimated)

PRIMARY OUTCOMES:
Assessment of excess body weight loss | 3 months after surgery
  During postoperative visits, the patient's body weight loss obtained after surgery will be assessed by means of absolute BMI values measured after the operative period and the percentage of lost BMI.
Assessment of excess body weight loss | 6 months after surgery
  During postoperative visits, the patient's body weight loss obtained after surgery will be assessed by means of absolute BMI values measured after the operative period and the percentage of lost BMI.
Assessment of excess body weight loss | 9 months after surgery
  During postoperative visits, the patient's body weight loss obtained after surgery will be assessed by means of absolute BMI values measured after the operative period and the percentage of lost BMI.
Assessment of excess body weight loss | 12 months after surgery
  During postoperative visits, the patient's body weight loss obtained after surgery will be assessed by means of absolute BMI values measured after the operative period and the percentage of lost BMI.
Assessment of excess body weight loss | 18 months after surgery
  During postoperative visits, the patient's body weight loss obtained after surgery will be assessed by means of absolute BMI values measured after the operative period and the percentage of lost BMI.
Assessment of the remaining stomach and duodenum access by endoscopy exam performed on each patient | 3 months after surgery
  To assess access to the remaining stomach and duodenum, endoscopies will be performed after surgery by a professional from the endoscopy team at Hospital Geral Alberto Rassi.
Assessment of the remaining stomach and duodenum access by endoscopy exam performed on each patient | 12 months after surgery
  To assess access to the remaining stomach and duodenum, endoscopies will be performed after surgery by a professional from the endoscopy team at Hospital Geral Alberto Rassi.
Assessment of the remaining stomach and duodenum access by endoscopy exam performed on each patient | 18 months after surgery
  To assess access to the remaining stomach and duodenum, endoscopies will be performed after surgery by a professional from the endoscopy team at Hospital Geral Alberto Rassi.
Application of the BAROS (Bariatric Analysis and Reporting Outcome) questionnaire | 6 months after surgery
  The questionnaire used for subjective evaluation of the surgery result and the post-operative quality of life adopted will be the BAROS (Bariatric Analysis and Reporting Outcome). The BAROS protocol consists of three major research areas (weight loss, medical conditions and quality of life questionnaire), from which a maximum score of three points is obtained for each category, totaling a maximum of nine points. The questionnaire will be applied by trained researchers.
Application of the BAROS (Bariatric Analysis and Reporting Outcome) questionnaire | 12 months after surgery
  The questionnaire used for subjective evaluation of the surgery result and the post-operative quality of life adopted will be the BAROS (Bariatric Analysis and Reporting Outcome). The BAROS protocol consists of three major research areas (weight loss, medical conditions and quality of life questionnaire), from which a maximum score of three points is obtained for each category, totaling a maximum of nine points. The questionnaire will be applied by trained researchers.
Application of the BAROS (Bariatric Analysis and Reporting Outcome) questionnaire | 18 months after surgery
  The questionnaire used for subjective evaluation of the surgery result and the post-operative quality of life adopted will be the BAROS (Bariatric Analysis and Reporting Outcome). The BAROS protocol consists of three major research areas (weight loss, medical conditions and quality of life questionnaire), from which a maximum score of three points is obtained for each category, totaling a maximum of nine points. The questionnaire will be applied by trained researchers.

SECONDARY OUTCOMES:
Weight loss assessment through exams and interviews | 18 months
  Monitoring of weight loss through weighing and questionnaire completed by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Reis Esselin de Melo, Principal Investigator — Hospital Geral de Goiânia
Locations (1):
- Paulo Reis Esselin de Melo, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No